CLINICAL TRIAL: NCT04537455
Title: Non-invasive Mapping Using Ultra-high Frequency Electrocardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19HH5155
Record Dates: First submitted 2020-08-28; First posted 2020-09-03 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Left Bundle-Branch Block; Right Bundle-Branch Block; Non-Specific Intraventricular Conduction Defect
Keywords: Ultra-high frequency electrocardiography; Left bundle branch block; Cardiac resynchronization Therapy; His Bundle Pacing
MeSH Terms: conditions — Bundle-Branch Block

STUDY DESIGN:
Intervention Model Description: Patients will have an ultra-high frequency electrocardiogram done.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abnormal cardiac conduction (Experimental): patients with abnormal cardiac conduction will undergo an ultra-high frequency electrocardiogram
  Interventions: Diagnostic Test: Ultra-high frequency electrocardiography

INTERVENTIONS:
Diagnostic Test: Ultra-high frequency electrocardiography — Patients will have an ultra-high frequency electrocardiography performed.

SUMMARY:
Cardiac electrical mapping is an important tool that allows doctors to study the electrical activity of the heart in detail. Electrical mapping systems used in clinical practice are time consuming, invasive and very costly. Ultra-high frequency electrocardiography is a novel non-invasive cardiac mapping system. Ultra-high frequency electrocardiography (UHF-ECG) can be performed in 10-15 minutes without any risk or discomfort to patients.

The aim of this study is to refine this mapping system, verify it against invasive mapping and develop software to bring this novel system into routine clinical use including predicting which patients will respond to cardiac resynchronisation therapy.

DETAILED DESCRIPTION:
This is a single centre laboratory study aiming to utilise ultra-high frequency electrocardiography to construct cardiac electrical activation maps.

All participants will attend for an UHF-ECG. This involves placing standard electrocardiography electrodes (up to 48) followed by electrocardiography recording using the UHF-ECG machine for 10-15 minutes.

Participants undergoing a clinically indicated VT ablation procedure will their UHF-ECG done before the procedure at a separate time. The ablation procedure itself will proceed as standard with no alternation whatsoever in study participants and no invasive measurements will be undertaken during the procedure. After the procedure is complete the 3D electrical maps collected to guide VT ablation will be analyzed and used for the study. The invasive maps will be compared with the non-invasive maps obtained using UHF-EGC.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age > 18 years)
* Able to give consent
* Some patients will be recruited from those listed for a clinically indicated VT ablation
* Patient subgroups as follows; 60 participants with LBBB undergoing a clinically indicated VT ablation , 20 participants with normal 12 lead ECG and normal left ventricular function assessed using standard echocardiography, 20 participants with right bundle branch block morphology on 12 lead ECG, 40 participants with non-specific conduction delay on 12 lead ECG, 60 participants with left bundle branch block morphology on 12 lead ECG and 20 participants who developed left bundle branch block morphology on 12 lead ECG after undergoing aortic valve replacement

Exclusion Criteria:

* Unable to give consent
* Children (age < 18 years)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Number of patients with block in the proximal conduction system | 3 years
  number of participant with an electrical activation map where the pattern indicates proximal conduction disease.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Whinnett, Study Director — Imperial College London
Locations (1):
- Hammersmith Hospital Imperial College NHS trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jurak P, Halamek J, Meluzin J, Plesinger F, Postranecka T, Lipoldova J, Novak M, Vondra V, Viscor I, Soukup L, Klimes P, Vesely P, Sumbera J, Zeman K, Asirvatham RS, Tri J, Asirvatham SJ, Leinveber P. Ventricular dyssynchrony assessment using ultra-high frequency ECG technique. J Interv Card Electrophysiol. 2017 Sep;49(3):245-254. doi: 10.1007/s10840-017-0268-0. Epub 2017 Jul 10. PMID 28695377